CLINICAL TRIAL: NCT04559269
Title: Micro-sleep During Maintenance Wakefulness Tests
Brief Title: Microsleep 1, Micro-sleep During Maintenance Wakefulness Tests
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2020_Microsleep1
Record Dates: First submitted 2020-07-02; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-07

CONDITIONS: Lobectomy; Hepatectomy; Pancreaticoduodenectomy
Keywords: Maintenance Wakefulness Tests; micro-sleep; sleepiness; latency; EEG
MeSH Terms: conditions — Sleepiness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Cohort of 98 patients suffering from sleep disorders hospitalized between September 2017 and January 2019 in the Sleep Medicine Center of the Croix Rousse Hospital (Lyon) for objective sleepiness evaluation with polysomnography and MWT.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — patients have benefited from maintenance wakefulness tests as part of their clinical evaluation

SUMMARY:
During general anesthesia, intraoperative hypotension (IOH) is associated with increased morbidity and mortality. Mean arterial pressure (MAP) < 65mmHg is the most common definition of hypotension. In order to reduce IOH, a complex method using machine learning called hypotensive prediction index (HPI) was shown to be superior to changes in MAP (ΔMAP) to predict hypotension (MAP between 65 and 75 excluded). Linear extrapolation of MAP (LepMAP) is also very simple and could be a better approach than ΔMAP. The main objective of the present study was to investigate whether LepMAP could predict IOH during anesthesia 1, 2 or 5 minutes before.

DETAILED DESCRIPTION:
Hypothesis : the area under the ROC curves (ROC AUCs) at 1, 2 and 5 minutes of LepMAP would be superior to AMAP

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from sleep pathologies (apneas, narcolepsy, etc.) hospitalized for polysomnography and MWT, in order to evaluate their sleepiness (usually before they resume driving)
* hospitalized in the Center for Sleep Medicine (Hôpital Lyon Croix Rousse) between September 2017 and January 2019

Exclusion Criteria:

* patient with active encephalopathy or epilepsy whose EEG was abnormal
* denial of study participation
* availability of all the recordings (n=4 tests) of the MWT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from sleep pathologies (apneas, narcolepsy, etc.) hospitalized for polysomnography and wakefulness tests, generally with a view to authorizing driving.
Sampling Method: Non-Probability Sample
Enrollment: 98 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
TThe primary endpoint was to determine if LepMAP was better than ΔMAP for the prediction of hypotensive event at 1, 2 and 5 minutes, defined as a mean arterial pressure of less than 65 mmHg | Only during perioperative period
  the number of patients with MS during MWT as well as the mean number of MS per patient will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital de la Croix Rousse / GHN, Lyon, France